CLINICAL TRIAL: NCT05027893
Title: Efficacy of the Application of Moxifloxacin and Cefixime in Reduction of Inflammatory Sequelae and Complications After Mandibular Third Molar Surgery
Brief Title: Complications After Lower Third Molar Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Branislav Bajkin, MD, DMD, PhD, University Full Professor, Vice Dean for PhD studies, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01-33/8-2019
Record Dates: First submitted 2021-07-27; First posted 2021-08-30 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Complications; Antibiotic Reaction; Antibiotic Side Effect; Antibiotic Resistant Infection; Antibiotic Resistant Strain; Infection, Bacterial; Infection, Laboratory
Keywords: Molar, Third; Moxifloxacin; Cefixime; Placebo; Postoperative Complications; Antibiotic Prophylaxis; Drug Resistance; Microbial Sensitivity Tests
MeSH Terms: conditions — Postoperative Complications; Bacterial Infections; Laboratory Infection | interventions — Moxifloxacin; Tablets; Cefixime

STUDY DESIGN:
Intervention Model Description: A RANDOMIZED CONTROLLED TRIAL
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients were randomly and equally assigned to treatment groups. The study was planned as a double-blind. Thus, neither the patients nor the researchers knew whether the patients were prescribed antibiotics or placebo tablets, because the tablets were marked with a label that was in the formed codebook. All the film-coated tablets used were of the same appearance (both the antibiotics and the placebo). There was 157 participants, patients and the same oral surgeon.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active Comparator: The first tested group (Active Comparator): Patients orally received film-coated tablets with either 400 mg of moxifloxacin. Film-coated tablets were administered for the first five days postoperatively, once a day, in a double-blind manner. All patients were evaluated at the postoperative follow-ups on the first, second and seventh postoperative day.
  Interventions: Drug: Moxifloxacin 400 mg Oral Tablet
- Active Comparator: The second tested group (Active Comparator): Patients orally received film-coated tablets with either 400 mg of cefixime. Film-coated tablets were administered for the first five days postoperatively, once a day, in a double-blind manner. All patients were evaluated at the postoperative follow-ups on the first, second and seventh postoperative day.
  Interventions: Drug: Cefixime 400 mg Oral Tablet
- Placebo Comparator: The control group (Placebo Comparator): One third of patients received placebo-tablets containing indifferent substances with no antimicrobial action (99% microcrystalline cellulose, 0.5% silicon dioxide and 0.5% magnesium stearate, which were of the same colour and overall appearance as the used antibiotics. Film-coated tablets were administered for the first five days postoperatively, once a day, in a double-blind manner. All patients were evaluated at the postoperative follow-ups on the first, second and seventh postoperative day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Moxifloxacin 400 mg Oral Tablet — All used film-coated tablets (400 mg moxifloxacin) were administered for the first five days postoperatively, once a day, after the lower third molar surgery.
  Other Names: perioperative/prophylaxis
  Arms: Active Comparator: The first tested group
Drug: Cefixime 400 mg Oral Tablet — All used film-coated tablets (400 mg cefixime) were administered for the first five days postoperatively, once a day, after the lower third molar surgery.
  Other Names: perioperative/prophylaxis
  Arms: Active Comparator: The second tested group
Other: Placebo — All used film-coated placebo-tablets were administered for the first five days postoperatively, once a day, after the lower third molar surgery.
  Arms: Placebo Comparator: The control group

SUMMARY:
Surgical removal of impacted mandibular wisdom teeth is a frequent intervention, usually accompanied by unpleasant sequelae (pain, swelling and trismus) in the postoperative period, sometimes even with possibly serious complications (dry socket/alveolar osteitis and postoperative infection at the surgical site - SSI). It is therefore advisable to use various medications and procedures to prevent or alleviate the occurrence of these sequelae and complications. Accordingly, there is a debate in the literature on the expedience of perioperative (prophylactic) use of antibiotics. It is interesting that numerous articles recommending perioperative (prophylactic) antibiotic use to patients undergoing the impacted mandibular third molar surgery may be found, as well as those providing arguments for the disagreement with such an approach, considering that its benefits do not outweigh the risks of adverse side effects, especially due to growing resistance of microorganisms towards antibiotics, which is a possible serious threat to global health. Concerning the perioperative (prophylactic) use of antibiotics for this indication, consensus has not yet been reached, and neither of the views has been verified by convincing scientific evidence. Having the aforementioned dilemma in mind, the main endpoint of the study was to determine the validity of perioperative (prophylactic) use of antibiotics as to alleviate customary sequelae and possible complications after surgical removal of impacted mandibular third molars and, at the same time, the effectiveness of newer antibiotics (moxifloxacin and cefixime) when used for this purpose. Moreover, microbiological investigations of susceptibility of the isolated microorganisms to antibiotics used in this research were performed, which could verify the clinically obtained results. With this in mind, two major contributions, based on scientifically verified results, could be expected from the research: (1) confirmation or refuting the validity of perioperative (prophylactic) antibiotic use to control sequelae or complications that could follow the impacted mandibular third molar surgery; and (2) confirmation of the efficacy of fluoroquinolones (moxifloxacin) and cephalosporins (cefixime) in controlling odontogenic infections.

DETAILED DESCRIPTION:
Clinical research was conducted at the Oral Surgery Department of the Dental Clinic of Vojvodina, Novi Sad, Serbia, adopting the double-blind prospective clinical study design. Microbiological studies were performed at the Center for Microbiology of the Institute of Public Health of Vojvodina, Novi Sad, Serbia, on swab samples obtained from the surgical wounds of patients with postoperative infection or the exudate (pus) obtained from the peri-coronal space of patients with pericoronitis or history of pericoronitis. The susceptibility of isolated microorganisms to moxifloxacin, cefixime and other antibiotics commonly used in oral & maxillofacial surgery (penicillin and its derivatives, erythromycin, azithromycin, clindamycin and tetracycline) was tested microbiologically. Patients ≥18 years, indicated for surgical removal of the impacted mandibular third molars, with good systemic health - patients classified as American Society of Anesthesiologists (ASA) classification of Physical Health is a grading system for preoperative health of the surgical patients - ASA I and ASA II were included in the study. Evaluation of the effects of the applied medication was performed on the basis of postoperative sequelae or complications. Complications, including dry socket/alveolar osteitis (AO) and postoperative infection at the surgical site (SSI), and inflammatory sequelae - pain, swelling and trismus (limited mouth opening), were evaluated postoperatively.

In the case of pericoronitis or a history of pericoronitis, with the presence of exudate or pus, as well as in the case of postoperative infection, a swab was taken from the operative wound or pericoronary space, and the punctate of exudate or pus was sent for microbiological analysis. The main goal of this analysis was to establish the susceptibility of microorganisms not only to antibiotics used in this study, but also to antibiotics, which are the "gold standard" in the treatment of odontogenic infections, as well as other commonly used antibiotics in the treatment. Analyses were performed by standard bacteriological techniques (seeding the material on appropriate nutrient media and incubating them at 35-37 °C for 18-24 h) to isolate the bacteria. Identification of bacterial species was performed by classical bacteriological methods (morphological, cultural and physiological-biochemical), as well as by the automated system Matrix Assisted Laser Desorption Ionization - Time of Flight (MALDI-TOF), Germany. After identification, susceptibility testing of isolated bacterial species to antimicrobial drugs was performed by standard disk-diffusion method according to Kirby-Bauer, Mueller-Hinton agar and blood Mueller-Hinton agar (HiMedia, India), depending on which bacterial species was in question in line with European Committee on Antimicrobial Susceptibility Testing (EUCAST) or Clinical & Laboratory Standards Institute (CLSI) Guidelines. Discs from Bio-Rad, France, were used to perform the microbiological analyses.

All surgical interventions were performed under local anesthesia, using 2% lidocaine with adrenaline 1: 80,000 in a total 4 ml volume (2 ml solution for injection contained 40 mg lidocaine hydrochloride in the form of lidocaine hydrochloride monohydrate and 0.025 mg adrenaline in the form of adrenaline tartrate: Lidocaine 2% - adrenaline, 40 mg +0.025. In all patients, the surgery involved a triangular mucoperiosteal flap design, sutured using synthetic poly-filament non-resorptive suture material (3-0). Patients were advised to take an analgesic containing 200 mg ibuprofen and 325 mg acetaminophen.

In accordance with known ethical principles and in accordance with the principles of Good Clinical Practice (GCP), care for the well-being of the patients was maximally respected, in accordance with the latest revision of the Declaration of Helsinki and accepted principles that apply to clinical trials on humans. The holder of the protection of the patients in this clinical trial was the principal researcher, who cooperated with the Ethics Committee of the Dental Clinic of Vojvodina, University of Novi Sad. The patients written Informed Consent implied that the patient had received full information about the research, and was stressed that they had the right to decide independently to participate, without coercion and external influences, or any harmful consequences if they refused to participate.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥18 years, indicated for surgical removal of the impacted mandibular third molars, with good systemic health (patients classified as ASA I and ASA II) were included in the study.

Exclusion Criteria:

* hypersensitivity to study drugs; history of systemic antibacterial therapy within 6 months prior to randomization; pregnancy or breastfeeding; fluoroquinolone-related tendon disorder; clinically relevant cardiac conditions or QT interval prolonging drugs; severe hepatic insufficiency (Child-Pugh C). Also, criteria for not including the patients in the study were cases where, in addition to removing the impacted mandibular third molar, some other oral surgical procedure was performed, as well as patients with currently present pericoronitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative infection at the surgical site (SSI) | Up to 12 weeks (3 months) after surgery.
  Signs of postoperative infection were registered clinically, based on the presence of local signs of inflammation and general signs of intoxication (elevated body temperature, accelerated erythrocyte sedimentation, leucocytosis, the level of C-reactive protein, etc. ).

SECONDARY OUTCOMES:
Dry socket (alveolar osteitis) | Through 7 days.
  The dry socket (alveolar osteitis) was diagnosed based on reported severe pain in the wound area, accompanied by specific local clinical appearance of the operative wound and absence of pus.
Postoperative pain assessed by visual analogue scale (VAS) | 1st, 2nd day and 7th day after surgery.
  The postoperative pain was assessed using a visual analogue scale (VAS). VAS represents a horizontally drawn length of 100 mm, the beginning of which indicates a pain-free state on the left side, and the end on the right side the state of the strongest pain imaginable. All patients, by placing a dash on the scale, indicated the intensity of pain that, on the appropriate day in the postoperative period, they felt in its strongest intensity. The intensity of pain was determined by measuring the distance of the marked place on the scale from the beginning of the scale on the left side and expressed in millimeters.
Postoperative swelling (oedema) | 1st, 2nd day and 7th day after surgery.
  The postoperative swelling (oedema) coefficient was obtained by measuring the preoperative and postoperative distance between specific reference points in millimetres. The reference points were: the outer corner of the eye and the angle of the lower jaw; lip corner and tragus; and chin tip and tragus.
Postoperative trismus (maximum inter-incisal opening of mouth) | 1st, 2nd day and 7th day after surgery.
  The degree of postoperative trismus was assessed by measuring the distance between mesio-incisal angles of the upper and lower central incisors at the maximum mouth opening ability.
Postoperative pain assessed by verbal rating scale (VRS) | 1st to 7th day after surgery.
  The postoperative pain was assessed using a verbal rating scale (VRS). VRS involves a numerical assessment of pain intensity based on six degrees (1-6) - no pain, barely sensitive pain, mild pain, moderate pain, severe pain and very strong, almost unbearable pain.
Postoperative pain assessed by number of analgesics | 1st to 7th day after surgery.
  In each patient, the moment of postoperative pain, its intensity at the indicated observation times was registered, and the need for additional analgesics was registered (patients recorded the number of analgesics consumed daily from the completed surgical intervention to suture removal in the postoperative pain monitoring protocol).

OTHER OUTCOMES:
Rate of antibiotic susceptibility and resistance of isolated microorganisms in vitro (microbiological assessment). | Up to 12 weeks (3 months) after surgery.
  The sensitivity of isolated microorganisms to moxifloxacin, cefixime and other antibiotics commonly prescribed in oral and maxillofacial surgery was tested microbiologically. Regarding the susceptibility to antimicrobial drugs, bacteria were classified according to the growth inhibition zone, into three categories: susceptible (S), intermediate (I) and resistant (R).
Incidence of adverse drug events (ADEs) in the clinical trial | Up to 24 days after surgery.
  During the study, any adverse event to drugs used in the clinical study will be recorded in accordance with the GCP.

CONTACTS AND LOCATIONS:
Overall Officials: Branislav V Bajkin, MD, DMD, PhD, Study Chair — Dental Clinic of Vojvodina, Faculty of Medicine, University of Novi Sad; Branimir D Stošić, DMD, PhD, Study Director — University of Novi Sad, Faculty of Medicine
Locations (1):
- Dental Clinic of Vojvodina, Faculty of Medicine, University of Novi Sad, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carter K, Worthington S. Predictors of Third Molar Impaction: A Systematic Review and Meta-analysis. J Dent Res. 2016 Mar;95(3):267-76. doi: 10.1177/0022034515615857. Epub 2015 Nov 11. PMID 26561441
- [Result] Bouloux GF, Steed MB, Perciaccante VJ. Complications of third molar surgery. Oral Maxillofac Surg Clin North Am. 2007 Feb;19(1):117-28, vii. doi: 10.1016/j.coms.2006.11.013. PMID 18088870
- [Result] Chuang SK, Perrott DH, Susarla SM, Dodson TB. Age as a risk factor for third molar surgery complications. J Oral Maxillofac Surg. 2007 Sep;65(9):1685-92. doi: 10.1016/j.joms.2007.04.019. PMID 17719384
- [Result] Azenha MR, Kato RB, Bueno RB, Neto PJ, Ribeiro MC. Accidents and complications associated to third molar surgeries performed by dentistry students. Oral Maxillofac Surg. 2014 Dec;18(4):459-64. doi: 10.1007/s10006-013-0439-9. Epub 2013 Dec 27. PMID 24370576
- [Result] Markovic AB, Todorovic L. Postoperative analgesia after lower third molar surgery: contribution of the use of long-acting local anesthetics, low-power laser, and diclofenac. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Nov;102(5):e4-8. doi: 10.1016/j.tripleo.2006.02.024. Epub 2006 Aug 10. PMID 17052624
- [Result] Schalch TO, Palmieri M, Longo PL, Braz-Silva PH, Tortamano IP, Michel-Crosato E, Mayer MPA, Jorge WA, Bussadori SK, Pavani C, Negreiros RM, Horliana ACRT. Evaluation of photodynamic therapy in pericoronitis: Protocol of randomized, controlled, double-blind study. Medicine (Baltimore). 2019 Apr;98(17):e15312. doi: 10.1097/MD.0000000000015312. PMID 31027098
- [Result] Kim JC, Choi SS, Wang SJ, Kim SG. Minor complications after mandibular third molar surgery: type, incidence, and possible prevention. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Aug;102(2):e4-11. doi: 10.1016/j.tripleo.2005.10.050. Epub 2006 Jun 27. PMID 16876044
- [Result] Monaco G, Staffolani C, Gatto MR, Checchi L. Antibiotic therapy in impacted third molar surgery. Eur J Oral Sci. 1999 Dec;107(6):437-41. doi: 10.1046/j.0909-8836.1999.eos107604.x. PMID 10625102
- [Result] Monaco G, Tavernese L, Agostini R, Marchetti C. Evaluation of antibiotic prophylaxis in reducing postoperative infection after mandibular third molar extraction in young patients. J Oral Maxillofac Surg. 2009 Jul;67(7):1467-72. doi: 10.1016/j.joms.2008.12.066. PMID 19531419
- [Result] Susarla SM, Dodson TB. Risk factors for third molar extraction difficulty. J Oral Maxillofac Surg. 2004 Nov;62(11):1363-71. doi: 10.1016/j.joms.2004.05.214. PMID 15510357
- [Result] Yuasa H, Kawai T, Sugiura M. Classification of surgical difficulty in extracting impacted third molars. Br J Oral Maxillofac Surg. 2002 Feb;40(1):26-31. doi: 10.1054/bjom.2001.0684. PMID 11883966
- [Result] Blum IR. Contemporary views on dry socket (alveolar osteitis): a clinical appraisal of standardization, aetiopathogenesis and management: a critical review. Int J Oral Maxillofac Surg. 2002 Jun;31(3):309-17. doi: 10.1054/ijom.2002.0263. PMID 12190139
- [Result] Bowe DC, Rogers S, Stassen LF. The management of dry socket/alveolar osteitis. J Ir Dent Assoc. 2011 Dec-2012 Jan;57(6):305-10. PMID 22338284
- [Result] Taberner-Vallverdu M, Nazir M, Sanchez-Garces MA, Gay-Escoda C. Efficacy of different methods used for dry socket management: A systematic review. Med Oral Patol Oral Cir Bucal. 2015 Sep 1;20(5):e633-9. doi: 10.4317/medoral.20589. PMID 26116842
- [Result] Taberner-Vallverdu M, Sanchez-Garces MA, Gay-Escoda C. Efficacy of different methods used for dry socket prevention and risk factor analysis: A systematic review. Med Oral Patol Oral Cir Bucal. 2017 Nov 1;22(6):e750-e758. doi: 10.4317/medoral.21705. PMID 29053647
- [Result] Kolokythas A, Olech E, Miloro M. Alveolar osteitis: a comprehensive review of concepts and controversies. Int J Dent. 2010;2010:249073. doi: 10.1155/2010/249073. Epub 2010 Jun 24. PMID 20652078
- [Result] Daly B, Sharif MO, Newton T, Jones K, Worthington HV. Local interventions for the management of alveolar osteitis (dry socket). Cochrane Database Syst Rev. 2012 Dec 12;12:CD006968. doi: 10.1002/14651858.CD006968.pub2. PMID 23235637
- [Result] Bortoluzzi MC, Capella DL, Barbieri T, Pagliarini M, Cavalieri T, Manfro R. A single dose of amoxicillin and dexamethasone for prevention of postoperative complications in third molar surgery: a randomized, double-blind, placebo controlled clinical trial. J Clin Med Res. 2013 Feb;5(1):26-33. doi: 10.4021/jocmr1160w. Epub 2013 Jan 11. PMID 23390473
- [Result] Ren YF, Malmstrom HS. Effectiveness of antibiotic prophylaxis in third molar surgery: a meta-analysis of randomized controlled clinical trials. J Oral Maxillofac Surg. 2007 Oct;65(10):1909-21. doi: 10.1016/j.joms.2007.03.004. PMID 17884515
- [Result] Benediktsdottir IS, Wenzel A, Petersen JK, Hintze H. Mandibular third molar removal: risk indicators for extended operation time, postoperative pain, and complications. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Apr;97(4):438-46. doi: 10.1016/j.tripleo.2003.10.018. PMID 15088029
- [Result] Blondeau F, Daniel NG. Extraction of impacted mandibular third molars: postoperative complications and their risk factors. J Can Dent Assoc. 2007 May;73(4):325. PMID 17484797
- [Result] Lodi G, Figini L, Sardella A, Carrassi A, Del Fabbro M, Furness S. Antibiotics to prevent complications following tooth extractions. Cochrane Database Syst Rev. 2012 Nov 14;11:CD003811. doi: 10.1002/14651858.CD003811.pub2. PMID 23152221
- [Result] Friedman JW. The prophylactic extraction of third molars: a public health hazard. Am J Public Health. 2007 Sep;97(9):1554-9. doi: 10.2105/AJPH.2006.100271. Epub 2007 Jul 31. PMID 17666691
- [Result] Salmeron-Escobar JI, del Amo-Fernandez de Velasco A. Antibiotic prophylaxis in Oral and Maxillofacial Surgery. Med Oral Patol Oral Cir Bucal. 2006 May 1;11(3):E292-6. PMID 16648771
- [Result] Rodrigues WC, Okamoto R, Pellizzer EP, dos Carrijo AC, de Almeida RS, de Melo WM. Antibiotic prophylaxis for third molar extraction in healthy patients: Current scientific evidence. Quintessence Int. 2015 Feb;46(2):149-61. doi: 10.3290/j.qi.a32825. PMID 25279397
- [Result] Moreno-Drada JA, Garcia-Perdomo HA. Effectiveness of Antimicrobial Prophylaxis in Preventing the Spread of Infection as a Result of Oral Procedures: A Systematic Review and Meta-Analysis. J Oral Maxillofac Surg. 2016 Jul;74(7):1313-21. doi: 10.1016/j.joms.2016.03.006. Epub 2016 Mar 15. PMID 27060492
- [Result] Moloney J, Stassen LF. Pericoronitis: treatment and a clinical dilemma. J Ir Dent Assoc. 2009 Aug-Sep;55(4):190-2. PMID 19753908
- [Result] Wehr C, Cruz G, Young S, Fakhouri WD. An Insight into Acute Pericoronitis and the Need for an Evidence-Based Standard of Care. Dent J (Basel). 2019 Sep 2;7(3):88. doi: 10.3390/dj7030088. PMID 31480662
- [Result] Davies SC, Fowler T, Watson J, Livermore DM, Walker D. Annual Report of the Chief Medical Officer: infection and the rise of antimicrobial resistance. Lancet. 2013 May 11;381(9878):1606-9. doi: 10.1016/S0140-6736(13)60604-2. Epub 2013 Mar 12. No abstract available. PMID 23489756
- [Result] Llor C, Bjerrum L. Antimicrobial resistance: risk associated with antibiotic overuse and initiatives to reduce the problem. Ther Adv Drug Saf. 2014 Dec;5(6):229-41. doi: 10.1177/2042098614554919. PMID 25436105
- [Result] Marra F, George D, Chong M, Sutherland S, Patrick DM. Antibiotic prescribing by dentists has increased: Why? J Am Dent Assoc. 2016 May;147(5):320-7. doi: 10.1016/j.adaj.2015.12.014. Epub 2016 Feb 5. PMID 26857041
- [Result] Roberts RM, Bartoces M, Thompson SE, Hicks LA. Antibiotic prescribing by general dentists in the United States, 2013. J Am Dent Assoc. 2017 Mar;148(3):172-178.e1. doi: 10.1016/j.adaj.2016.11.020. Epub 2017 Jan 23. PMID 28126225
- [Result] Palmer NA, Pealing R, Ireland RS, Martin MV. A study of therapeutic antibiotic prescribing in National Health Service general dental practice in England. Br Dent J. 2000 May 27;188(10):554-8. doi: 10.1038/sj.bdj.4800538. PMID 10870281
- [Result] Loffler C, Bohmer F, Hornung A, Lang H, Burmeister U, Podbielski A, Wollny A, Kundt G, Altiner A. Dental care resistance prevention and antibiotic prescribing modification-the cluster-randomised controlled DREAM trial. Implement Sci. 2014 Feb 22;9:27. doi: 10.1186/1748-5908-9-27. PMID 24559212
- [Result] Loffler C, Bohmer F. The effect of interventions aiming to optimise the prescription of antibiotics in dental care-A systematic review. PLoS One. 2017 Nov 14;12(11):e0188061. doi: 10.1371/journal.pone.0188061. eCollection 2017. PMID 29136646
- [Result] Wilson W, Taubert KA, Gewitz M, Lockhart PB, Baddour LM, Levison M, Bolger A, Cabell CH, Takahashi M, Baltimore RS, Newburger JW, Strom BL, Tani LY, Gerber M, Bonow RO, Pallasch T, Shulman ST, Rowley AH, Burns JC, Ferrieri P, Gardner T, Goff D, Durack DT; American Heart Association. Prevention of infective endocarditis: guidelines from the American Heart Association: a guideline from the American Heart Association Rheumatic Fever, Endocarditis and Kawasaki Disease Committee, Council on Cardiovascular Disease in the Young, and the Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and the Quality of Care and Outcomes Research Interdisciplinary Working Group. J Am Dent Assoc. 2008 Jan;139 Suppl:3S-24S. doi: 10.14219/jada.archive.2008.0346. PMID 18167394
- [Result] Dayer MJ, Jones S, Prendergast B, Baddour LM, Lockhart PB, Thornhill MH. Incidence of infective endocarditis in England, 2000-13: a secular trend, interrupted time-series analysis. Lancet. 2015 Mar 28;385(9974):1219-28. doi: 10.1016/S0140-6736(14)62007-9. Epub 2014 Nov 18. PMID 25467569
- [Result] Richey R, Wray D, Stokes T; Guideline Development Group. Prophylaxis against infective endocarditis: summary of NICE guidance. BMJ. 2008 Apr 5;336(7647):770-1. doi: 10.1136/bmj.39510.423148.AD. No abstract available. PMID 18390528
- [Result] Diz Dios P, Tomas Carmona I, Limeres Posse J, Medina Henriquez J, Fernandez Feijoo J, Alvarez Fernandez M. Comparative efficacies of amoxicillin, clindamycin, and moxifloxacin in prevention of bacteremia following dental extractions. Antimicrob Agents Chemother. 2006 Sep;50(9):2996-3002. doi: 10.1128/AAC.01550-05. PMID 16940094
- [Result] Limeres J, Sanroman JF, Tomas I, Diz P. Patients' perception of recovery after third molar surgery following postoperative treatment with moxifloxacin versus amoxicillin and clavulanic acid: a randomized, double-blind, controlled study. J Oral Maxillofac Surg. 2009 Feb;67(2):286-91. doi: 10.1016/j.joms.2008.06.061. PMID 19138601
- [Result] Cervino G, Cicciu M, Biondi A, Bocchieri S, Herford AS, Laino L, Fiorillo L. Antibiotic Prophylaxis on Third Molar Extraction: Systematic Review of Recent Data. Antibiotics (Basel). 2019 May 2;8(2):53. doi: 10.3390/antibiotics8020053. PMID 31052566
- [Result] Sidana S, Mistry Y, Gandevivala A, Motwani N. Evaluation of the Need for Antibiotic Prophylaxis During Routine Intra-alveolar Dental Extractions in Healthy Patients: A Randomized Double-Blind Controlled Trial. J Evid Based Dent Pract. 2017 Sep;17(3):184-189. doi: 10.1016/j.jebdp.2017.04.007. Epub 2017 Apr 27. PMID 28865815
- [Result] Prajapati A, Prajapati A, Sathaye S. Benefits of not Prescribing Prophylactic Antibiotics After Third Molar Surgery. J Maxillofac Oral Surg. 2016 Jun;15(2):217-20. doi: 10.1007/s12663-015-0814-1. Epub 2015 Jul 5. PMID 27298545
- [Result] Kaczmarzyk T, Wichlinski J, Stypulkowska J, Zaleska M, Panas M, Woron J. Single-dose and multi-dose clindamycin therapy fails to demonstrate efficacy in preventing infectious and inflammatory complications in third molar surgery. Int J Oral Maxillofac Surg. 2007 May;36(5):417-22. doi: 10.1016/j.ijom.2006.12.003. Epub 2007 Apr 3. PMID 17408924
- [Result] Marcussen KB, Laulund AS, Jorgensen HL, Pinholt EM. A Systematic Review on Effect of Single-Dose Preoperative Antibiotics at Surgical Osteotomy Extraction of Lower Third Molars. J Oral Maxillofac Surg. 2016 Apr;74(4):693-703. doi: 10.1016/j.joms.2015.11.017. Epub 2015 Nov 23. PMID 26706491
- [Result] Lopez-Cedrun JL, Pijoan JI, Fernandez S, Santamaria J, Hernandez G. Efficacy of amoxicillin treatment in preventing postoperative complications in patients undergoing third molar surgery: a prospective, randomized, double-blind controlled study. J Oral Maxillofac Surg. 2011 Jun;69(6):e5-14. doi: 10.1016/j.joms.2011.01.019. Epub 2011 Apr 5. PMID 21470751
- [Result] Halpern LR, Dodson TB. Does prophylactic administration of systemic antibiotics prevent postoperative inflammatory complications after third molar surgery? J Oral Maxillofac Surg. 2007 Feb;65(2):177-85. doi: 10.1016/j.joms.2006.10.016. PMID 17236918
- [Result] Arteagoitia I, Diez A, Barbier L, Santamaria G, Santamaria J. Efficacy of amoxicillin/clavulanic acid in preventing infectious and inflammatory complications following impacted mandibular third molar extraction. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Jul;100(1):e11-8. doi: 10.1016/j.tripleo.2005.03.025. PMID 15953905
- [Result] Menon RK, Gopinath D, Li KY, Leung YY, Botelho MG. Does the use of amoxicillin/amoxicillin-clavulanic acid in third molar surgery reduce the risk of postoperative infection? A systematic review with meta-analysis. Int J Oral Maxillofac Surg. 2019 Feb;48(2):263-273. doi: 10.1016/j.ijom.2018.08.002. Epub 2018 Aug 23. PMID 30145064
- [Result] Pham TDM, Ziora ZM, Blaskovich MAT. Quinolone antibiotics. Medchemcomm. 2019 Jun 28;10(10):1719-1739. doi: 10.1039/c9md00120d. eCollection 2019 Oct 1. PMID 31803393
- [Result] Ardila CM, Guzman IC. Clinical Factors Influencing the Efficacy of Systemic Moxifloxacin in the Therapy of Patients With Generalized Aggressive Periodontitis: A Multilevel Analysis From a Clinical Trial. Glob J Health Sci. 2015 Jun 25;8(3):80-8. doi: 10.5539/gjhs.v8n3p80. PMID 26493435
- [Result] Sobottka I, Wegscheider K, Balzer L, Boger RH, Hallier O, Giersdorf I, Streichert T, Haddad M, Platzer U, Cachovan G. Microbiological analysis of a prospective, randomized, double-blind trial comparing moxifloxacin and clindamycin in the treatment of odontogenic infiltrates and abscesses. Antimicrob Agents Chemother. 2012 May;56(5):2565-9. doi: 10.1128/AAC.06428-11. Epub 2012 Feb 21. PMID 22354306
- [Result] Shrivastava R, Rai VK, Kumar A, Sinha S, Tripathi P, Gupta K, Sabharwal S. An in vitro Comparison of Endodontic Medicaments Propolis and Calcium Hydroxide alone and in Combination with Ciprofloxacin and Moxifloxacin against Enterococcus Faecalis. J Contemp Dent Pract. 2015 May 1;16(5):394-9. doi: 10.5005/jp-journals-10024-1696. PMID 26162260
- [Result] Jones ME, Visser MR, Klootwijk M, Heisig P, Verhoef J, Schmitz FJ. Comparative activities of clinafloxacin, grepafloxacin, levofloxacin, moxifloxacin, ofloxacin, sparfloxacin, and trovafloxacin and nonquinolones linozelid, quinupristin-dalfopristin, gentamicin, and vancomycin against clinical isolates of ciprofloxacin-resistant and -susceptible Staphylococcus aureus strains. Antimicrob Agents Chemother. 1999 Feb;43(2):421-3. doi: 10.1128/AAC.43.2.421. PMID 9925551
- [Result] Dalhoff A. Immunomodulatory activities of fluoroquinolones. Infection. 2005 Dec;33 Suppl 2:55-70. doi: 10.1007/s15010-005-8209-8. PMID 16518713
- [Result] Dalhoff A, Shalit I. Immunomodulatory effects of quinolones. Lancet Infect Dis. 2003 Jun;3(6):359-71. doi: 10.1016/s1473-3099(03)00658-3. PMID 12781508
- [Result] Lang MS, Gonzalez ML, Dodson TB. Do Antibiotics Decrease the Risk of Inflammatory Complications After Third Molar Removal in Community Practices? J Oral Maxillofac Surg. 2017 Feb;75(2):249-255. doi: 10.1016/j.joms.2016.09.044. Epub 2016 Oct 6. PMID 28341449
- [Result] Ardila CM, Florez-Florez J, Castaneda-Parra LD, Guzman IC, Bedoya-Garcia JA. Moxifloxacin versus amoxicillin plus metronidazole as adjunctive therapy for generalized aggressive periodontitis: a pilot randomized controlled clinical trial. Quintessence Int. 2020;51(8):612-621. doi: 10.3290/j.qi.a44715. PMID 32507863
- [Result] Oomens MA, Forouzanfar T. Antibiotic prophylaxis in third molar surgery: a review. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Dec;114(6):e5-12. doi: 10.1016/j.oooo.2011.10.023. Epub 2012 May 30. PMID 23159124
- [Result] Poeschl PW, Eckel D, Poeschl E. Postoperative prophylactic antibiotic treatment in third molar surgery--a necessity? J Oral Maxillofac Surg. 2004 Jan;62(1):3-8; discussion 9. doi: 10.1016/j.joms.2003.05.004. PMID 14699540
- [Result] Warnke PH, Becker ST, Springer IN, Haerle F, Ullmann U, Russo PA, Wiltfang J, Fickenscher H, Schubert S. Penicillin compared with other advanced broad spectrum antibiotics regarding antibacterial activity against oral pathogens isolated from odontogenic abscesses. J Craniomaxillofac Surg. 2008 Dec;36(8):462-7. doi: 10.1016/j.jcms.2008.07.001. Epub 2008 Aug 29. PMID 18760616
- [Result] Tally FP, Desjardins RE, McCarthy EF, Cartwright K. Safety profile of cefixime. Pediatr Infect Dis J. 1987 Oct;6(10):976-80. doi: 10.1097/00006454-198710000-00037. PMID 3320926
- [Result] Martens E, Demain AL. The antibiotic resistance crisis, with a focus on the United States. J Antibiot (Tokyo). 2017 May;70(5):520-526. doi: 10.1038/ja.2017.30. Epub 2017 Mar 1. PMID 28246379
- [Result] Lacasa JM, Jimenez JA, Ferras V, Bossom M, Sola-Morales O, Garcia-Rey C, Aguilar L, Garau J. Prophylaxis versus pre-emptive treatment for infective and inflammatory complications of surgical third molar removal: a randomized, double-blind, placebo-controlled, clinical trial with sustained release amoxicillin/clavulanic acid (1000/62.5 mg). Int J Oral Maxillofac Surg. 2007 Apr;36(4):321-7. doi: 10.1016/j.ijom.2006.11.007. Epub 2007 Jan 16. PMID 17229548
- [Result] Blumenthal KG, Lu N, Zhang Y, Walensky RP, Choi HK. Recorded Penicillin Allergy and Risk of Mortality: a Population-Based Matched Cohort Study. J Gen Intern Med. 2019 Sep;34(9):1685-1687. doi: 10.1007/s11606-019-04991-y. No abstract available. PMID 31011962
- [Result] Redgrave LS, Sutton SB, Webber MA, Piddock LJ. Fluoroquinolone resistance: mechanisms, impact on bacteria, and role in evolutionary success. Trends Microbiol. 2014 Aug;22(8):438-45. doi: 10.1016/j.tim.2014.04.007. Epub 2014 May 16. PMID 24842194
- [Result] Chaudhry SB, Veve MP, Wagner JL. Cephalosporins: A Focus on Side Chains and beta-Lactam Cross-Reactivity. Pharmacy (Basel). 2019 Jul 29;7(3):103. doi: 10.3390/pharmacy7030103. PMID 31362351
- [Result] Al-Nawas B, Walter C, Morbach T, Seitner N, Siegel E, Maeurer M, Krummenauer F. Clinical and microbiological efficacy of moxifloxacin versus amoxicillin/clavulanic acid in severe odontogenic abscesses: a pilot study. Eur J Clin Microbiol Infect Dis. 2009 Jan;28(1):75-82. doi: 10.1007/s10096-008-0587-2. Epub 2008 Jul 29. PMID 18663500
- [Result] Nymoen Aasbrenn M, Skeie I, Berild D. Compliance to antibiotic guidelines leads to more appropriate use of antibiotics in skin and soft tissue infections in injecting drug users. Infect Dis (Lond). 2019 Aug;51(8):570-577. doi: 10.1080/23744235.2019.1617435. Epub 2019 May 30. PMID 31144548
- [Result] Poeschl PW, Spusta L, Russmueller G, Seemann R, Hirschl A, Poeschl E, Klug C, Ewers R. Antibiotic susceptibility and resistance of the odontogenic microbiological spectrum and its clinical impact on severe deep space head and neck infections. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Aug;110(2):151-6. doi: 10.1016/j.tripleo.2009.12.039. Epub 2010 Mar 25. PMID 20346713
- [Result] Arteagoitia MI, Barbier L, Santamaria J, Santamaria G, Ramos E. Efficacy of amoxicillin and amoxicillin/clavulanic acid in the prevention of infection and dry socket after third molar extraction. A systematic review and meta-analysis. Med Oral Patol Oral Cir Bucal. 2016 Jul 1;21(4):e494-504. doi: 10.4317/medoral.21139. PMID 26946211
- [Result] Gomez-Arambula H, Hidalgo-Hurtado A, Rodriguez-Flores R, Gonzalez-Amaro AM, Garrocho-Rangel A, Pozos-Guillen A. Moxifloxacin versus Clindamycin/Ceftriaxone in the management of odontogenic maxillofacial infectious processes: A preliminary, intrahospital, controlled clinical trial. J Clin Exp Dent. 2015 Dec 1;7(5):e634-9. doi: 10.4317/jced.52627. eCollection 2015 Dec. PMID 26644841
- [Result] Daabiss M. American Society of Anaesthesiologists physical status classification. Indian J Anaesth. 2011 Mar;55(2):111-5. doi: 10.4103/0019-5049.79879. PMID 21712864
- See also: A comparative analysis of the efficacy of moxifloxacin and cefixime in reduction postoperative inflammatory sequelae after mandibular third molar surgery — http://www.doiserbia.nb.rs/Article.aspx?id=0042-84502000122S#.YPhwrtUzaM8